CLINICAL TRIAL: NCT04730687
Title: Er,Cr:YSGG and Diode Lasers in the Treatment of Peri-implantitis: A Randomized Clinical Trial
Brief Title: Er,Cr:YSGG and Diode Lasers in the Treatment of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nazli Zeynep Alpaslan Yayli, PhD, DDA, Assistant professor, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21.11.2018/02
Record Dates: First submitted 2021-01-19; First posted 2021-01-29 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Peri-Implantitis
Keywords: Peri-implant disease; laser therapy; Er,Cr:YSGG; Diode; MMP-9; TIMP-1
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional non-surgical mechanical therapy (Placebo Comparator): Mechanical instrumentation in all groups continued with titanium Gracey curettes (8mm in diameter, Langer ½, item code: 7103, Kohler Medizintechnik, GmbH & Co, Ltd, Stockach, Germany) until the clinician gently felt that the surface was sufficiently debrided.There is no laser application. The laser tip is placed in the peri-implant sulcus but not activated.
  Interventions: Device: Traditional non surgical mechanical therapy
- Diode laser-assisted non-surgical mechanical therapy (Active Comparator): 1 week after mechanical debridment, 940 nm diode laser (Ezlase®, Biolase Technology, Inc., San Clemente, CA) has been applied with the aid of a 300 µm diameter optical fiber tip (E3-9 mm) placed approximately 1 mm above the most apical part of the peri implant pocket, parallel to the implant surface. Pocket irrigation was performed with 3% hydrogen peroxide solution for 10 seconds before and after diode laser application.The fiber was moved in apico-coronal and mesial-distal directions for a total of 30 seconds during laser light emission.The laser tip was checked every 7-8 seconds and wiped with sterile saline in order to prevent a possible coagulation or temperature increase.The laser was used in continuous pulse mode, at a power of 0.8 Watt (W), an energy density of 3J / cm2 and a spot diameter of 1 mm. Pulse width and pulse interval were applied as 20 milliseconds.
  Interventions: Device: Diode laser assisted non-surgical mechancal therapy
- Er, Cr: YSGG laser-assisted non-surgical mechanical therapy (Active Comparator): 1 week after mechanical debridment, 2780 nm Er, Cr: YSGG laser (Waterlase®, Biolase Technology, Inc., San Clemente, CA), with 500 µm diameter fiberoptic periodontal tip (RFPT5-14 mm) was applied in short pulse '' H '' mode, water cooled with a non-contact sweeping motion for 30 seconds parallel to the implant surface.The settings used are: 1.5 W power, 30 Hz frequency, 50% water, 40% air, 140 s pulse duration and 1 cm spot size.
  Interventions: Device: Er, Cr: YSGG laser-assisted non-surgical mechanical therapy

INTERVENTIONS:
Device: Traditional non surgical mechanical therapy — Mechanical instrumentation in all groups was made with titanium Gracey curettes (8mm in diameter, Langer ½, item code: 7103, Kohler Medizintechnik, GmbH & Co, Ltd, Stockach, Germany).
  Arms: Traditional non-surgical mechanical therapy
Device: Diode laser assisted non-surgical mechancal therapy — One week after mechanical treatment, a 940 nm diode laser (Ezlase®, Biolase Technology, Inc., San Clemente, CA) with a 300 µm diameter optical fiber tip applied approximately 1 mm above the most apical part of the peri-implant pocket, parallel to the implant surface (E3-9 mm).
  Arms: Diode laser-assisted non-surgical mechanical therapy
Device: Er, Cr: YSGG laser-assisted non-surgical mechanical therapy — 1 week after mechanical treatment, 2780 nm Er, Cr: YSGG laser (Waterlase®, Biolase Technology, Inc., San Clemente, CA), short pulse '' H '' with 500 µm diameter fiberoptic periodontal tip (RFPT5-14 mm) mode has been applied.
  Arms: Er, Cr: YSGG laser-assisted non-surgical mechanical therapy

SUMMARY:
In this study, 940 nm diode laser and 2780 nm erbium, chromium doped: yttrium, scandium, gallium, garnet (Er, Cr: YSGG) laser were used in the non-surgical treatment of peri-implant diseases in addition to mechanical treatment. And the effects of dental lasers on clinical parameters and matrix metalloproteinase 9 (MMP-9) and tissue inhibitors of matrix metalloproteinases-1 (TIMP-1) levels in peri-implant crevicular fluid were evaluated.

DETAILED DESCRIPTION:
With the widespread use of dental implants, there is an increase in technical and biological complications. These complications are called peri-implant diseases in general terms. When peri-implant diseases are not treated, a process that progresses to the loss of the affected implant may develop, but there is still no accepted consensus on their treatment.When performing treatment procedures, it is recommended not only to remove inflamed tissues but also to decontaminate infected implant surfaces.Recently, with the development of laser technologies, the use of dental lasers in implant surface detoxification has come to the fore. Dental lasers attract increasing attention due to their anti-infective properties, easy handling and haemostatic effects against periodontal pathogens.Diode lasers attract attention with their safety when used directly on the implant surface, soft tissue penetration, antibacterial and biostimulating properties. They detoxify implant surfaces by killing pathogenic bacteria through photothermal effects and neutralizing bacterial endotoxins. Erbium lasers also show promising results in implant treatment due to their advantageous properties such as soft and hard tissue ablation and decontamination. Er, Cr: YSGG lasers have the ability to debride microstructured surfaces of dental implants without causing mechanical damage, thanks to their ability to work with water.Today, many researchers investigate the effectiveness of dental lasers in the treatment of peri-implant diseases, but it has not yet been proven whether they have an additional contribution. It is observed that studies mostly focus on clinical parameters. However, it is stated that periodontal probing and radiographs, which are used as common diagnostic methods, may give erroneous results. These methods refer only to pre-existing destruction rather than current disease activity. A model predicting the course of peri-implant disease has not yet been defined, but biomarkers may offer considerable potential for disease activity.Biomarkers are widely used in medicine to objectively determine disease state or responses to a therapeutic intervention. Gingival fluid (GCF) biomarkers have moderate diagnostic validity in periodontitis. It is stated that biomarkers in peri-implant groove fluid (PICF) also give promising results in terms of diagnosis and prognostic values. MMP-8 and MMP-9, the two main collagen degrading enzymes in GCF, are secreted from neutrophils during disease activation and are responsible for extracellular matrix degradation. TIMP-1, a major inhibitor of MMPs, has been reported to be released at high levels in inflamed gums.

In the literature review, it has been observed that there are quite a limited number of human clinical studies investigating the effect of dental lasers of different wavelengths on treatment results in the treatment of peri-implant disease at the clinical and molecular level. The aim of this study is to investigate the effects of 940 nm diode laser and 2780 nm Er, Cr: YSGG laser-assisted non-surgical mechanical treatment on clinical parameters and MMP-9 and TIMP-1 levels in PICF in individuals with peri-implant disease.

ELIGIBILITY:
Inclusion Criteria:

1. Inflammation in the peri-implant area,

   1. Probing depth ≥ 3 mm in one or more areas,
   2. Bleeding with probing with or without suppuration under light forces (0.25 N)
   3. Patients with bone loss [Patients with bone loss ≥ 2mm identified as peri-implantitis],
2. There is no evidence of occlusal overload,
3. Implant-supported fixed prosthesis that has been in use for at least 6 months in the mouth and does not interfere with the evaluation of clinical parameters.

Exclusion Criteria:

1. Smoking
2. Having a systemic disease that may affect the treatment results such as uncontrolled diabetes, metabolic bone diseases, hematological disorders, radiotherapy in the head and neck region, kidney disease,
3. Being in pregnancy or breastfeeding period,
4. Using antibiotics and / or non-steroidal anti-inflammatory drugs in the last 3 months,
5. Steroid and bisphosphonate use,
6. To have any dental treatment in the last 3 months,
7. Requiring surgical techniques in the treatment of peri-implant disease.

Ages: 35 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Plaque index score (0-3) | 6 months
  Plaque index was measured from the 4 surfaces of each implant. The plaque index score of each implant was calculated with Silness-Loe plaque index by dividing the total value by 4.
  0:absence of microbial plaque
  1. Thin film of microbial plaque along the free peri-implant margin
  2. moderate accumulation with plaque in the sulcus
  3. large amount of plaque in sulcus or pocket along the free peri-implant margin
Gingival index score (0-3) | 6 months
  The gingival index was measured from the 4 surfaces of each implant. The gingival index score of each implant was calculated with Silness-Loe gingival indeks by dividing the total value by 4.
  0:Normal gingiva
  1. Mild inflammation: slight change in color, slight oedema, no bleeding on probing
  2. Moderate inflammation: redness,oedema and glazing, bleeding on probing
  3. Severe inflammation: marked redness and oedema, ulceration, tendency to spontaneous bleeding
Bleeding on probing (percentage) | 6 months
  Bleeding on probing was measured by Ainamo and Bay's gingival bleeding index from 4 surfaces of each implant. If there is bleeding after probing, it is recorded as +, if there is no bleeding it is recorded as _. Gingival bleeding index is calculated as a percentage of affected sites.
Probing depth (mm) | 6 months
  Probing depth (PD) (distance from peri-implant margin to peri-implant pocket base) was measured with a plastic probe (UNC 12 Colorvue probe, Hu-Friedy, Chicago, USA) in 4 regions (mesial, buccal, distal, lingual / palatinal) of each implant and recorded as mm.
Matrix Metalloproteinase-9 (MMP-9) level (ng/mL) | 6 months
  Samples were collected using specially prepared paper strips (PerioPaper, Oraflow, NY, USA). The strips were stored in 1.5 mL sterile eppendorf tubes with 500μl phosphate-based saline (PBS) at pH 7.4. and -40 ° C. PICF samples were collected again from the same site of the same implant at 6 months following the treatments. When the targeted number is reached, in the investigation of MMP-9 levels in PICF, enzyme-linked immunosorbent assay (ELISA) is carried out in line with the recommendations of the manufacturer (Human Matrix Metalloproteinase-9 ELISA Kit, Bioassay Technology Laboratory, Shanghai, China). Absorbance values were read with a 450 nm wavelength ELISA reader (µQuantTM ELISA Microplate Reader, BioTek® Instruments, Inc., Vermont, USA).
Tissue Inhibitors of Metalloproteinase-1 (TIMP-1) level (pg/mL) | 6 months
  Samples were collected using specially prepared paper strips (PerioPaper, Oraflow, NY, USA). The strips were stored in 1.5 mL sterile eppendorf tubes with 500μl phosphate-based saline (PBS) at pH 7.4. and -40 ° C. PICF samples were collected again from the same site of the same implant at 6 months following the treatments. When the targeted number is reached, in the investigation of TIMP-1 levels in PICF, enzyme-linked immunosorbent assay (ELISA) is carried out in line with the recommendations of the manufacturer (Human Tissue Inhibitors of Metalloproteinase-1 ELISA Kit, Bioassay Technology Laboratory, Shanghai, China). Absorbance values were read with a 450 nm wavelength ELISA reader (µQuantTM ELISA Microplate Reader, BioTek® Instruments, Inc., Vermont, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Nazli Zeynep Alpaslan Yayli, PhD, Principal Investigator — Yuzuncu Yil University; Ahmet Cemil Talmac, PhD, Study Chair — Yuzuncu Yil University; Serap Keskin Tunc, PhD, Study Chair — Yuzuncu Yil University; Damla Akbal, PhD, Study Chair — Yuzuncu Yil University; Dicle Altindal, PhD, Study Chair — Yuzuncu Yil University; Abdullah Seckin Ertugrul, Professor, Study Chair — Izmir Katip Celebi University
Locations (1):
- Nazli Zeynep Alpaslan Yayli, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sinjab K, Garaicoa-Pazmino C, Wang HL. Decision Making for Management of Periimplant Diseases. Implant Dent. 2018 Jun;27(3):276-281. doi: 10.1097/ID.0000000000000775. PMID 29762186
- [Derived] Alpaslan Yayli NZ, Talmac AC, Keskin Tunc S, Akbal D, Altindal D, Ertugrul AS. Erbium, chromium-doped: yttrium, scandium, gallium, garnet and diode lasers in the treatment of peri-implantitis: clinical and biochemical outcomes in a randomized-controlled clinical trial. Lasers Med Sci. 2022 Feb;37(1):665-674. doi: 10.1007/s10103-021-03436-5. Epub 2021 Oct 12. PMID 34637055